CLINICAL TRIAL: NCT05273528
Title: A Single Arm, Open Label Clinical Study to Evaluate the Immunogenicity and Safety of Sequential Immunization of V-01-351/V-01D Bivalence Vaccine in Healthy Adults Aged 18 Years and Older After the Vaccination of 2 Doses of Inactivated Vaccines
Brief Title: The Immunogenicity and Safety of V-01-351/V-01D Bivalence Vaccine
Acronym: Omicron
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V-01-351/V-01D-Booster-02
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V-01-351/V-01D bivalence vaccine (Experimental)
  Interventions: Biological: Recombinant SARS-CoV-2 Beta Variant Fusion Protein Vaccine/Recombinant SARS-CoV-2 Delta Variant Fusion Protein Vaccine

INTERVENTIONS:
Biological: Recombinant SARS-CoV-2 Beta Variant Fusion Protein Vaccine/Recombinant SARS-CoV-2 Delta Variant Fusion Protein Vaccine — The product should be a milky-white suspension for injection. For prevention of SARS-CoV-2 infection.
  Other Names: V-01-351/V-01D Bivalence Vaccine

SUMMARY:
It is a Single Arm, Open Label Clinical Study to Evaluate the Immunogenicity and Safety of Sequential Immunization of V-01-351/V-01D Bivalence Vaccine in Healthy Adults Aged 18 Years and Older After the Vaccination of 2 Doses of Inactivated Vaccines. A total of 20 participants were enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants aged 18 years and older who have completed the second dose of 2-dose regimen of SARS-CoV-2 vaccine (Vero cell) Inactivated in the past 4-8 months;
2. Voluntarily participate in the study and sign the informed consent form, who can provide valid ID and follow the study protocol requirement;
3. In the past 14 days, no history of high or medium risk of the epidemic, overseas travel history or residence history; no history of contact with confirmed, asymptomatic or suspected COVID-19 cases; no history of contact with the persons from high- and medium-risk epidemic areas or contact patients with fever or respiratory symptoms; and those who are not in isolation period.
4. Males of reproductive potential and females of childbearing potential voluntarily agree to take effective and acceptable contraceptive methods from the signing of informed consent form to 3 months after vaccination.

Exclusion Criteria:

1. Confirmed COVID-19 cases, or positive for SARS-CoV-2 test by RT-PCR. 2. History of previous SARS infection. 3. History of severe allergy to any vaccine or any ingredient of the vaccine including aluminum adjuvant, e.g., anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction), dyspnea, angioedema, etc..

4. People who currently suffer from the following diseases:

1. Symptoms related to acute respiratory infections (such as: sneezing, nasal congestion, runny nose, cough, sore throat, loss of taste, chills, shortness of breath, etc.)
2. Patients with thrombocytopenia, any coagulation dysfunction, or receive anticoagulant treatment, etc.
3. Patients with congenital or acquired angioedema/neuroedema;
4. A history of congenital or acquired immunodeficiency or autoimmune disease (except for mild psoriasis, controllable autoimmune thyroid disease, vitiligo, or stable celiac disease that does not require immunosuppressive or immunomodulatory therapy); no spleen , or history of spleen surgery, history of trauma, or treatment with immunomodulators within 6 months, such as: glucocorticoid with the dose causing immunosuppressive (dose reference: equivalent to prednisone 20mg/day, more than one week); or monoclonal antibody ; or thymosin; or interferon, etc.; but local medication (such as ointment, eye drops, inhalation or nasal spray) is allowed.
5. Patients with active tuberculosis, viral hepatitis, human immunodeficiency virus or syphilis infection.
6. Patients with acute diseases, or acute attacks of chronic diseases, or uncontrolled severe chronic diseases: history of chronic respiratory diseases (including moderate to severe asthma, COPD, pulmonary fibrosis), hypertension that cannot be controlled by drugs (systolic blood pressure ≥150mmHg) And/or diastolic blood pressure ≥100mmHg), history of severe cardiovascular disease (including heart failure, coronary artery disease, cardiomyopathy), history of chronic kidney disease, history of cancer (except for basal cell carcinoma), diabetes (unsatisfied blood sugar control or diabetes related serious complications).

5. Received attenuated live vaccine within 28 days before the vaccination or any subunit vaccines and inactivated vaccines within 14 days before the vaccination.

6. Injection of immunoglobulin and/or other blood products within 3 months before the administration of study vaccine; or with the plan to use such product within 6 month after immunization.

7. Pregnant (including positive urine pregnancy test for women of childbearing age) or breastfeeding women. Or women or their partners who have a pregnancy plan within 3 months after the trial vaccination.

8. Have participated in or are participating in other COVID-19 related clinical trials, or are participating in other drug clinical trials; 9. Those considered by the investigator as inappropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2023-01-06 (Estimated); Study Completion 2023-01-06 (Estimated)

PRIMARY OUTCOMES:
GMT of neutralizing antibody | 28 days after booster immunization
  GMT of neutralizing antibody (pesudovirus/live virus) of SARS-CoV-2 Omicron variant after 14 days and 28 days administered with V-01-351/V-01D Bivalence Vaccine
GMI of neutralizing antibody | 28 days after booster immunization
  GMI of neutralizing antibody (pesudovirus/live virus) of SARS-CoV-2 Omicron variant after 14 days and 28 days administered with V-01-351/V-01D Bivalence Vaccine
Seroconversion rate of neutralizing antibody | 28 days after booster immunization
  Seroconversion rate of neutralizing antibody (pesudovirus/live virus) of SARS-CoV-2 Omicron variant after 14 days and 28 days administered with V-01-351/V-01D Bivalence Vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- Shaoguan Hospital of Chinese Medicine, Shaoguan, Guangdong, China